CLINICAL TRIAL: NCT02668757
Title: Pilot Study, How the HeartHab Application Can Support Coronary Artery Disease Patients in Their Rehabilitation Program?
Brief Title: HeartHab, Can a Patient-tailored Application Support Coronary Artery Disease Patients During Rehabilitation?
Acronym: HeartHab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HeartHab-001
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HeartHab application arm (Other): Patients in the HeartHab application arm will receive the mobile application during study period.
  Interventions: Behavioral: HeartHab application intervention

INTERVENTIONS:
Behavioral: HeartHab application intervention — The intervention patients will use the HeartHab application on a smartphone. During the study, the patients will use the HeartHab application for 4-6 weeks.

SUMMARY:
The HeartHab study is a pilot trial in which coronary artery disease patients (n = 15-30) are given the HeartHab application. The HeartHab application is a smarthphone based mobile application that serves as a secondary prevention tool, to support cardiac patients after their phase II cardiac rehabilitation program. During study period (4-6 weeks), participating patients will be asked to use the application. HeartHab includes a module devoted to therapy compliance, one to exercise training prescription and one to risk factor control. HeartHab aims to motivate the patient to improve his/her self-management skills and hence decrease cardiovascular morbidity (and mortality).

Motivational aspects and usability data will be collected during study period by means of app logs and/or questionnaires/interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease for which they received a percutaneous coronary intervention, coronary artery bypass grafting or drugs only.
* Patients that have completed the standard cardiac rehabilitation program
* Patients who have access to a computer and a WiFi internet connection
* Patients that are able to go to the rehabilitation centre ReGo of Jessa Hospital
* Patients who signed the informed consent document

Exclusion Criteria:

* Patients with a history of VF, sustained VT and/or supraventricular tachycardia during the last 6 months before enrollment.
* Patients who due to cognitive, neurological and/or musculoskeletal constraints are unable to ride a bicycle.
* Patients with a pacemaker or defibrillator.
* Non-Dutch speaking patients
* Patients who simultaneously participate in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Impact on motivation | week 6
  By means of a questionnaire and an interview, questions are asked about participants' motivation for a tour

SECONDARY OUTCOMES:
Usability of the HeartHab application | week 6
  By means of a questionnaire and an interview, the participants are asked about the usability of the application. This information will give insights in parts of the application that could be improved considering the usability

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, Prof. dr., Principal Investigator — paul.dendale@jessazh.be
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No